CLINICAL TRIAL: NCT03509272
Title: LimPrOn: Limburg Pre-eclampsia Investigation
Acronym: LimPrOn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Wilfried Gyselaers, Principal Investigator, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Limpron-001
Record Dates: First submitted 2016-08-24; First posted 2018-04-26 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy; Pre-eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention)
- remote monitoring group (Experimental)
  Interventions: Device: remote monitoring

INTERVENTIONS:
Device: remote monitoring — Intervention Description: Patients can participate in the study when they're 10 weeks pregnant. At 10 weeks: a NICCOMO, Maternal Venous Doppler Echography and Maltron measurement will be taken. This measurement will be repeated at 20 weeks of pregnancy, and 30 weeks of pregnancy when they're aberrant.
  When the measurements are abnormal, the patients will be included in the remote monitoring study. The following protocol and devices will be applied:
  Device What When Withings Wireless Blood Pressure Monitor Blood Pressure 2x/day Withings Pulse O² Activity Day and night Withings Smart Body Analyzer Weight
  1x/day
  Arms: remote monitoring group

SUMMARY:
Background:

Multiple adaptations at the cardiovascular system occurs during pregnancy. In the pregnancy condition pre-eclampsia (PE), this adaptations are abnormal. Five to eight percent of all pregnant women worldwide will develop PE.

PE is a pregnancy condition which is characterized with a high blood pressure (>140/90 mm Hg) and the occurrence of proteinuria (>3g/dl/24h) after 20 weeks of gestation. When untreated, this condition can have severe complications for both mother and child. It's important to monitor women with a high risk for developing PE for an early detection and treatment of this condition.

For this reason, a multicenter study is set up with the following applications:

1. NICCOMO and Maternal Venous Doppler Echography: impedance cardiograph and an echography of the heart and veins.
2. Maltron: bio-electronic impedance analyze
3. Remote monitoring of the high risk patients to become a more intensive follow-up

Number of inclusions: 2000 pregnant women from the prenatal consultations of eight different hospitals:

ELIGIBILITY:
Inclusion Criteria:

* > 10 weeks of pregnancy, primipara and multipara

Exclusion Criteria:

* < 10 weeks of pregnancy and congenital malformations of the fetus

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2016-05; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Niccomo measurement | 10 weeks of pregnancy
  The NICOMMO can record can record multiple haemodynamic parameters uninterrupted and reliable in an objective manner by using Impedance Cardiography. This technology is simple and non-invasive, and safe for pregnant women. The aim of this course is to describe the course of these parameters through normal pregnancies, and to examine any abnormalities in pre-eclamptic pregnancies. In view of the fact that in pre-eclampsia certain cardiovascular parameters are abnormal during several weeks before the disease becomes clinically manifest, this device might have a potential role in the prediction of pre-eclampsia in the future.
Niccomo measurement | 20 weeks of pregnancy
  The NICOMMO can record can record multiple haemodynamic parameters uninterrupted and reliable in an objective manner by using Impedance Cardiography. This technology is simple and non-invasive, and safe for pregnant women. The aim of this course is to describe the course of these parameters through normal pregnancies, and to examine any abnormalities in pre-eclamptic pregnancies. In view of the fact that in pre-eclampsia certain cardiovascular parameters are abnormal during several weeks before the disease becomes clinically manifest, this device might have a potential role in the prediction of pre-eclampsia in the future.
Systolic and Diastolic Blood pressure monitoring | 10 weeks of pregnancy
Systolic and Diastolic Blood pressure monitoring | 20 weeks of pregnancy
a maternal Venous Doppler Echochraphy | 10 weeks of pregnancy
  In cardiology, a combined ultrasound ECG study provides important information about the functioning of the heart, especially with regard to the "stiffening" of the heart and blood vessel walls. It is known that in pre-eclampsia the blood vessel walls stiffen. Up to now it has never been investigated whether a combined Echo-ECG study can provide information about the degree of vascular wall stiffening. This study component checks which reference values are in normal pregnancy and whether these differ from pre-eclamptic pregnancies.
Maltron measurement | 10 weeks of pregnancy
  The aim of this course is to describe the course of body composition and fluid balance through a normal pregnancy, and to examine any abnormalities in pre-eclamptic pregnancies.
a maternal Venous Doppler Echochraphy | 20 weeks of pregnancy
  In cardiology, a combined ultrasound ECG study provides important information about the functioning of the heart, especially with regard to the "stiffening" of the heart and blood vessel walls. It is known that in pre-eclampsia the blood vessel walls stiffen. Up to now it has never been investigated whether a combined Echo-ECG study can provide information about the degree of vascular wall stiffening. This study component checks which reference values are in normal pregnancy and whether these differ from pre-eclamptic pregnancies.
Maltron measurement | 20 weeks of pregnancy
  The aim of this course is to describe the course of body composition and fluid balance through a normal pregnancy, and to examine any abnormalities in pre-eclamptic pregnancies.
Activity tracker | 10 weeks of pregnancy
  Activity (amount of steps) will be checked to see if there is any correlation between the total amount of steps per day and the development of gestational hypertensive disorders.
Weight | 10 weeks of pregnancy
Activity tracker | 20 weeks of pregnancy
  Activity (amount of steps) will be checked to see if there is any correlation between the total amount of steps per day and the development of gestational hypertensive disorders.
Weight | 20 weeks of pregnancy

SECONDARY OUTCOMES:
birth weight | up to six weeks after delivery
gestational age | at the moment of delivery
  These data will be measured at the moment of delivery
mode of delivery | at the moment of delivery
intentioned start of delivery | at the moment of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Gyselaers, prof. dr., Principal Investigator — Hasselt University; Nele Geusens, dr., Study Chair — Ziekenhuis Oost-Limburg
Locations (8):
- Belgium (8):
  - Ziekenhuis Maas en Kempen, Bree
  - Ziekenhuis Oost-Limburg, Genk
  - Jessa Ziekenhuis, Hasselt
  - Sint-Fransiscus Ziekenhuis, Heusden-Zolder
  - Heilig Hart Ziekenhuis, Mol
  - Mariaziekenhuis Oost-Limburg, Overpelt
  - Sint-Trudo ziekenhuis, Sint-Truiden
  - AZ-vesalius, Tongeren

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394
- [Derived] Vandenberk T, Lanssens D, Storms V, Thijs IM, Bamelis L, Grieten L, Gyselaers W, Tang E, Luyten P. Relationship Between Adherence to Remote Monitoring and Patient Characteristics: Observational Study in Women With Pregnancy-Induced Hypertension. JMIR Mhealth Uhealth. 2019 Aug 28;7(8):e12574. doi: 10.2196/12574. PMID 31464190